CLINICAL TRIAL: NCT02611479
Title: Understanding Non-Response in Spine Fusion Surgery
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, David Flum, Medical Director, Surgical Outcomes Research Center, University of Washington
Other Study IDs: STUDY00001700; R21AR068009 (NIH)
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Results first posted 2019-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Spine Fusion
Keywords: patient reported outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To identify patient characteristics associated with non-response after spine fusion surgery for the treatment of degenerative disc disease (DDD).

ELIGIBILITY:
Inclusion Criteria:

* Subject has diagnosis of degenerative disc disease
* Subject is undergoing lumbar spine fusion surgery

Exclusion Criteria:

* Subject is less than 18 years of age
* Subject is not fluent in English
* Subject requires a caretaker for medical decision making

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (18 and over) undergoing spine fusion surgery in Washington State.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy M Cizik, MPH, PhC, Study Director — University of Washington
Locations (4):
- United States (4):
  - University of Washington, Seattle, Washington
  - Proliance Surgeons, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - Confluence Health, Wenatchee, Washington

REFERENCES:
- See also: Related Info — http://www.becertain.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: If participants did not complete a baseline survey before their lumbar spine fusion surgery or were found to be ineligible they were excluded from the study before completing follow-up surveys.
Groups:
- Spine Fusion Participants: Patients undergoing lumbar spine fusion surgery for any indication.
Period: Baseline Enrollment
Arm/Group | Spine Fusion Participants
Started | 184
Completed | 171
Not Completed | 13
Not completed — Exited study | 13
Period: Post-Surgery Follow-up at 30-90 Days
Arm/Group | Spine Fusion Participants
Started | 171
Completed | 169
Not Completed | 2
Not completed — No surgery reported | 2
Period: Post-Surgery Follow-up at 1-Year
Arm/Group | Spine Fusion Participants
Started | 169
Completed | 151
Not Completed | 18
Not completed — Lost to Follow-up | 18
Period: Data Cleaning
Arm/Group | Spine Fusion Participants
Started | 151
Completed | 149
Not Completed | 2
Not completed — No baseline function or pain metrics | 2

BASELINE CHARACTERISTICS:
Arm/Group | Spine Fusion Participants
Number analyzed (Participants) | 149
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 71
  >=65 years | 78
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There is 1 missing.
  Participants
    number analyzed (Participants) | 148
    Female | 83
    Male | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 144
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 140
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 149
Functional Limitations from back pain (ODI) [Mean (Standard Deviation); unit: units on a scale] — Oswestry Low Back Pain Disability Index (ODI) Total Score Scale 0-100 Sub-Scale Measures (0-5) for each: pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, and traveling.
  Interpretation: Simply add up your points for each section and plug it in to the following formula in order to calculate your level of disability: point total / 50 X 100 = % disability (aka: 'point total' divided by '50' multiply by ' 100 = percent disability)
  Lower values represent better outcomes. Higher values represent worse outcomes.
  units on a scale | 41.3 (15.4)
Anxiety [Mean (Standard Deviation); unit: T-scores] — PROMIS T Score: Total Anxiety Score 4 questions scaled 1-5 about anxiety, the raw score is the sum of these questions
  Formula: (Raw sum x number of items on the short form)/Number of items that were actually answered
  The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Therefore a person with a T-score of 40 is one SD below the mean. The standardized T-score is reported as the final score for each participant.
  Lower values represent better outcomes. Higher values represent worse outcomes.
  T-scores | 55.0 (9.2)
Depression [Mean (Standard Deviation); unit: T-scores] — PROMIS T Score: Total Depression Score 4 questions scaled 1-5 about depression, the raw score is the sum of these questions
  Formula: (Raw sum x number of items on the short form)/Number of items that were actually answered
  The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Therefore a person with a T-score of 40 is one SD below the mean. The standardized T-score is reported as the final score for each participant.
  Lower values represent better outcomes. Higher values represent worse outcomes.
  T-scores | 52.5 (9.6)
Sleep [Mean (Standard Deviation); unit: T-scores] — PROMIS T Score: Total Sleep Disturbance Score 4 questions scaled 1-5 about sleep disturbance, the raw score is the sum of these questions
  Formula: (Raw sum x number of items on the short form)/Number of items that were actually answered
  The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Therefore a person with a T-score of 40 is one SD below the mean. The standardized T-score is reported as the final score for each participant.
  Lower values represent worse outcomes. Higher values represent better outcomes.
  T-scores | 55.4 (7.4)
Pain chronicity [Count of Participants; unit: Participants]
  1-3 months | 1
  3-6 months | 4
  6 months-1 year | 19
  1-5 years | 39
  More than 5 years | 51
  Missing | 35
Pain interference [Mean (Standard Deviation); unit: T-scores] — PROMIS T Score: Total Pain Interference Score 4 questions scaled 1-5 about pain interference, the raw score is the sum of these questions
  Formula: (Raw sum x number of items on the short form)/Number of items that were actually answered
  The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Therefore a person with a T-score of 40 is one SD below the mean. The standardized T-score is reported as the final score for each participant.
  Lower values represent better outcomes. Higher values represent worse outcomes.
  T-scores | 67.1 (5.5)
Pain catastrophizing (fear avoidance) [Count of Participants; unit: Participants]
  Not at all | 30
  To a slight degree | 38
  To a moderate degree | 38
  To a great degree | 28
  All the time | 11
Alcohol, Marijuana Use [Count of Participants; unit: Participants]
  Alcohol | 42
  Cannabis Use: Score Recoded | 27
  Missing | 80
Asthma [Count of Participants; unit: Participants]
  No | 106
  Yes | 37
  Missing | 6
Opioid/additional therapies use [Count of Participants; unit: Participants] | 88
Global health [Count of Participants; unit: Participants] — PROMIS G02: general quality of life
  Participants
    Poor | 9
    Fair | 43
    Good | 61
    Very good | 28
    Excellent | 8
Emotional support [Mean (Standard Deviation); unit: T-scores] — PROMIS T Score: Total Emotional Support Score 4 questions scaled 1-5 about emotional support, the raw score is the sum of these questions
  Formula: (Raw sum x number of items on the short form)/Number of items that were actually answered
  The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Therefore a person with a T-score of 40 is one SD below the mean. The standardized T-score is reported as the final score for each participant.
  Lower values represent better outcomes. Higher values represent worse outcomes.
  T-scores | 54.8 (8.1)
Instrumental support [Mean (Standard Deviation); unit: T-scores] — PROMIS T Score: Total Instrumental Support Score 4 questions scaled 1-5 about instrumental support, the raw score is the sum of these questions
  Formula: (Raw sum x number of items on the short form)/Number of items that were actually answered
  The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Therefore a person with a T-score of 40 is one SD below the mean. The standardized T-score is reported as the final score for each participant.
  Lower values represent better outcomes. Higher values represent worse outcomes.
  T-scores | 55.2 (8.8)
Radiculopathy [Count of Participants; unit: Participants] | 112

OUTCOME MEASURES:

1. Primary Outcome: Oswestry Disability Index
Description: Change in pain and function after spine fusion surgery was measured by the Oswestry Disability Index. Scores range from 0 to 100.
  The questionnaire has 10 questions about pain intensity, personal care, lifting ability, walking ability, sitting ability, standing ability, sleeping ability, sex ability, social life, and travelling. Each question is followed by 6 options which describe the amount of disability a patient may face in these situations and the patient marks the statement most applicable to them. Each question is scored on a scale (0-5) with the first option "0" indicating the least amount of disability and "5" indicating the most severe disability. Higher scores indicate worse outcomes, lower scores indicate better outcomes.
Time Frame: Baseline, 60 day, 1 year
Population: 140 participants out of the 149 baseline participant population were analyzed since 9 participants were excluded due to incomplete Oswestry Disability Index data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Spine Fusion Participants
Number analyzed (Participants) | 140
score on a scale
  Baseline | 41.3 (15.4)
  60-day | 30.4 (17.1)
  12-month | 19.4 (17.3)

ADVERSE EVENTS:
Time Frame: Adverse Events not tracked and are inapplicable to this study.
Description: Adverse Events not tracked and are inapplicable to this study.
Arm/Group | Spine Fusion Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Clinical variables were collected from SCOAP which is a quality improvement database and variables are not as reliable as research variables. It is unknown if participants that did not complete the surveys would have responded to surgery or not.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/79/NCT02611479/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/79/NCT02611479/SAP_001.pdf